CLINICAL TRIAL: NCT01220739
Title: Safety of Rt-PA + Transcranial Emission of Low-Energy Lasers for Acute Stroke Recovery
Acronym: StELLAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Device sponsor no longer in business.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Justin Zivin, Professor, Department of Neurosciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StELLAR; P50NS044148 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; transcranial laser; tissue plasminogen activator; therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV tPA + Sham Transcranial Laser Therapy (Sham Comparator): Subjects in this treatment arm will receive IV tPA within 3 hours of stroke symptom onset followed by sham transcranial laser therapy no sooner than 12 hours after tPA and no greater than 24 hours from stroke onset.
  Interventions: Device: Transcranial Laser Therapy
- IV tPA +Transcranial Laser Therapy (Active Comparator): Subjects in this treatment arm will receive IV tPA within 3 hours of stroke symptom onset followed by transcranial laser therapy no sooner than 12 hours after tPA and no greater than 24 hours from stroke onset.
  Interventions: Device: Transcranial Laser Therapy

INTERVENTIONS:
Device: Transcranial Laser Therapy — Transcranial laser therapy is administered with the NeuroThera® Laser System (NTS) in subjects diagnosed with acute ischemic stroke. A laser system is a medical instrument that concentrates energy light on an area. Laser treatment has been used to deliver intense light energy to aid in the healing of tissues and wounds. The transcranial laser treatment procedure consists of applying the NTS laser to twenty different sites on the skull for two minutes at each site.
  Other Names: TLT; NeuroThera Laser System (NTS)

SUMMARY:
To assess the safety and preliminary efficacy of combining intravenous rt-PA with transcranial laser therapy (TLT) with the NeuroThera® Laser System (referred to hereafter as NTS) in subjects treated for acute ischemic stroke. Treatment with IV rt-PA must begin within 3 hours of symptom onset, and the initiation of TLT procedure must be feasible for each subject within 6 hours of stroke onset. The NeuroThera® Laser System is an investigational device that provides noninvasive transcranial laser therapy to subjects diagnosed with acute ischemic stroke. The wavelength of the laser light is in the infrared zone of the electromagnetic spectrum and is invisible to the naked eye.

DETAILED DESCRIPTION:
This study is a phase II (n= 200), prospective, double-blind, randomized, sham-controlled, multicenter, safety study of intravenous (IV) rt-PA alone versus IV rt-PA plus TLT (Transcranial Laser Therapy) at approximately 10 investigational sites (United States only). The primary endpoint for this safety study is occurrence of symptomatic intracranial hemorrhages at 36 - 48 hours after stroke symptom onset.

Symptomatic hemorrhage will be defined as deterioration of more than 4 points on the NIHSS lasting at least 72 hours accompanied by intracranial hemorrhage in the distribution of the neurological deficit as identified by neuroimaging scans. All follow up neuroimaging scans will be reviewed centrally by an independent reviewer for the presence or absence of hemorrhage on the 36-48 hour scan.

The secondary endpoints for this study are as follows:

* Hemorrhagic transformation without clinical consequences (asymptomatic) within 36-48 hours. All follow-up neuroimaging scans will be reviewed centrally by an independent reviewer for the presence or absence of hemorrhage on the 36-48 hour scan.
* Mortality
* The modified Rankin Scale (mRS) score dichotomized as 0-1 versus an mRS score of 2-6 at 90 days or the last rating in patients that develop intracerebral hemorrhages
* Frequency of SAEs and AEs This study is a phase II (N = 200), prospective, double-blind, randomized, sham controlled, multicenter, safety study of intravenous (IV) tissue plasminogen activator (rt-PA) versus IV rt-PA plus transcranial laser therapy (TLT) at approximately 10 investigational sites.

The study population will be randomized into two arms. One group will receive a sham TLT procedure (Sham Control Group or SCG) and the second group will receive an active TLT procedure (TLTG).

The randomization ratio of SCG and TLTG will be 1:1 and will be stratified in order to ensure balanced subject distribution between the treatment and sham-controlled groups for the following factors:

* Stroke severity as measured by National Institute of Health Stroke Scale (NIHSS) at baseline (stratified as 7-9, 10-13, 14-17)
* Study Site There are 6 visits in the study. The purpose of the Visit 1 will be to determine and confirm the eligibility of patients for participation in the StELLAR Study and document baseline information about the subject and their stroke event. This will include all of the following standard of care tests and procedures: a non contrast head CT scan performed prior to rt-PA administration, vital signs, height , weight ,physical exam, finger stick or blood glucose, serum or urine pregnancy test (if women of childbearing potential). In addition, the following data will be obtained: prestroke mRS, NIHSS, presumed location of stroke and vascular territory, start and stop date and time of the IV rt-PA treatment and dose given, date and time of stroke onset, date and time of arrival to the hospital, demographic data (date of birth, gender, ethnicity),sociodemographic data (education, marital status, social support prior to stroke),medical and surgical history (specific cardiovascular, neurological, endocrine, and other standard questions asked), method of contraception use (for women of child bearing potential), prior (three days prior to Screening) and current concomitant medication use, smoking history, adverse events from the time of obtaining informed consent. To be eligible for the study, the administration of rt-PA should follow the guidelines outlined by the National Institutes of Neurologic Disorders. Patients meeting the inclusion/exclusion criteria will be enrolled into the study after written informed consent is obtained by the patient or their legally authorized representative.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study only if they meet all of the following criteria:

1. Subject is at least 40 years of age at screening, but has not had their 81st birthday.
2. Subject has received IV rt-PA per the NINDS rt-PA Protocol Guidelines within 3 hours of symptom onset for an acute ischemic stroke.
3. Subject is diagnosed with acute ischemic stroke and presents to the health care facility at a time such that initiation of NTS procedure is feasible within 6 hours of the time of stroke onset. The time of stroke onset is defined as the time at which a change in the baseline neurological function occurred. If the time is not known (e.g., the subject awakens from sleep with new symptoms), the last time the patient was observed to be neurologically intact must be considered to be the time of onset.
4. Documented baseline NIHSS score of > 7 and < 17 prior to IV rt-PA administration. Subjects who transfer from other facilities after receiving IV rt-PA must have a documented NIHSS by a certified examiner prior to initiation of rt-PA treatment. Documentation of NIHSS score via telemedicine is acceptable if performed by a certified examiner. Subjects who improve prior to NTS procedure will still be treated, unless their NIHSS improves to 0.
5. Full functional independence just prior to the present stroke episode as defined by the following criteria:

   * Estimated prestroke mRS score 0 or 1.
   * Ambulates independently, may need a cane or walker, but does not need the assistance of another person.
   * Absence of a medical/physical/mental condition that substantially limits the subject's ability to work, study, participate in leisure activities, or look after family at home
   * Completely independent, does not need supervision (may live with other individuals, but could live alone if necessary)
6. Negative serum or urine pregnancy test in females of childbearing potential.
7. Subject (or legally authorized representative) provides written Informed Consent in compliance with local regulations prior to enrollment into this study.
8. The subject (and caregiver, if applicable) is willing to participate in this study for at least 90 days after the onset of stroke.-

Exclusion Criteria:

1. Evidence on from a pre-tPA head CT of an intracranial, subdural, or subarachnoid hemorrhage or clinical presentation suggestive of subarachnoid hemorrhage even if the initial neuroimaging scan is normal.
2. Clinical presentation consistent with a brainstem or cerebellar stroke
3. A rapidly improving neurological status that in the opinion of the investigator will make the subject unsuitable for participation in this study or patient rapidly improves to NIHSS of 0 by start of NTS procedure.
4. The subject had a seizure at stroke onset or within the 7 days prior to stroke onset.
5. Sustained blood glucose > 300 mg/dl or < 60 mg/dl
6. Subjects who, on repeated measurement, have a systolic blood pressure > 185, or a diastolic blood pressure > 110mmHg, post rt-PA administration, or it is the opinion of the investigator that aggressive treatment to reduce blood pressure post thrombolysis is required to keep pressure within these limits.
7. Presumed and/or confirmed septic embolus.
8. The subject has a history of CNS vascular wall disease (e.g. aneurysm, AVM).
9. The subject has a history of CNS disease or damage (e.g. neoplasm or dementia) which may influence the subject's outcome assessment.
10. The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on their scalp that is found to be directly below three or more TLT procedure sites.
11. Planned or actual use of any intra-arterial thrombolytic medication or a clot retrieval device, or any diagnostic or therapeutic interventional neurovascular procedure, including mechanical recanalization, whether successful or unsuccessful, during this stroke episode.
12. Subject previously participated in another investigational drug or device trial within the preceding four weeks.
13. Subject is a female who is pregnant or lactating (within the previous 30 days),or who is of child-bearing potential unless she is surgically sterile or she and/or her partner are using a medically acceptable method of birth control.
14. The subject has an implant of any kind in the head (i.e. clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
15. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.
16. The subject participated in the NEST-1, NEST-2, or NEST-3 Study.
17. The subject has any co-existing or terminal disease that may limit life expectancy or any medical condition (e.g. morbid obesity, substance abuse) that may, in the clinical judgment of the Investigator, independently influence the subject's outcome during the course of the study.
18. The subject is otherwise determined, based on the opinion of the Investigator,to be an unsuitable candidate for enrollment in this study. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hemmen, MD, PhD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - Swedish Medical Center, Englewood, Colorado
  - Palmetto Health Richland, Columbia, South Carolina
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the NINDS data sharing website.

REFERENCES:
- [Background] Zivin JA, Albers GW, Bornstein N, Chippendale T, Dahlof B, Devlin T, Fisher M, Hacke W, Holt W, Ilic S, Kasner S, Lew R, Nash M, Perez J, Rymer M, Schellinger P, Schneider D, Schwab S, Veltkamp R, Walker M, Streeter J; NeuroThera Effectiveness and Safety Trial-2 Investigators. Effectiveness and safety of transcranial laser therapy for acute ischemic stroke. Stroke. 2009 Apr;40(4):1359-64. doi: 10.1161/STROKEAHA.109.547547. Epub 2009 Feb 20. PMID 19233936
- [Background] Hacke W, Schellinger PD, Albers GW, Bornstein NM, Dahlof BL, Fulton R, Kasner SE, Shuaib A, Richieri SP, Dilly SG, Zivin J, Lees KR; NEST 3 Committees and Investigators. Transcranial laser therapy in acute stroke treatment: results of neurothera effectiveness and safety trial 3, a phase III clinical end point device trial. Stroke. 2014 Nov;45(11):3187-93. doi: 10.1161/STROKEAHA.114.005795. Epub 2014 Oct 7. PMID 25293665
- [Background] Huisa BN, Stemer AB, Walker MG, Rapp K, Meyer BC, Zivin JA; NEST-1 and -2 investigators. Transcranial laser therapy for acute ischemic stroke: a pooled analysis of NEST-1 and NEST-2. Int J Stroke. 2013 Jul;8(5):315-20. doi: 10.1111/j.1747-4949.2011.00754.x. Epub 2012 Feb 2. PMID 22299818

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Transcranial Laser Therapy: Subjects in this treatment arm will receive IV tPA within 3 hours of stroke symptom onset followed by sham transcranial laser therapy no sooner than 12 hours after tPA and no greater than 24 hours from stroke onset.
  Transcranial Laser Therapy: Transcranial laser therapy is administered with the NeuroThera® Laser System (NTS) in subjects diagnosed with acute ischemic stroke. A laser system is a medical instrument that concentrates energy light on an area. Laser treatment has been used to deliver intense light energy to aid in the healing of tissues and wounds. The transcranial laser treatment procedure consists of applying the NTS laser to twenty different sites on the skull for two minutes at each site.
- Transcranial Laser Therapy: Subjects in this treatment arm will receive IV tPA within 3 hours of stroke symptom onset followed by transcranial laser therapy no sooner than 12 hours after tPA and no greater than 24 hours from stroke onset.
  Transcranial Laser Therapy: Transcranial laser therapy is administered with the NeuroThera® Laser System (NTS) in subjects diagnosed with acute ischemic stroke. A laser system is a medical instrument that concentrates energy light on an area. Laser treatment has been used to deliver intense light energy to aid in the healing of tissues and wounds. The transcranial laser treatment procedure consists of applying the NTS laser to twenty different sites on the skull for two minutes at each site.
Period: Overall Study
Arm/Group | Sham Transcranial Laser Therapy | Transcranial Laser Therapy
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Transcranial Laser Therapy | Transcranial Laser Therapy | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.5) | 66.8 (12.7) | 65.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 3 | 7
Randomization NIH Stroke Scale [Mean (Standard Deviation); unit: score on a scale] — Total score is reported. Minimum score = 0 (better outcome); Maximum score = 42 (worse outcome)
  score on a scale | 12.3 (3.2) | 15.0 (2.4) | 13.4 (3.1)
Post-tPA Baseline/Treatment NIH Stroke Scale [Mean (Standard Deviation); unit: score on a scale] — Total score is reported. Minimum score = 0 (better outcome); Maximum score = 42 (worse outcome)
  score on a scale | 8.7 (5.4) | 9.6 (5.4) | 9.1 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Intracranial Hemorrhages
Time Frame: 36 hours from tPA initiation
Measure: Number; unit: participants
Arm/Group | Sham Transcranial Laser Therapy | Transcranial Laser Therapy
Number analyzed (Participants) | 7 | 5
participants | 0 | 0

2. Primary Outcome: Percentage of Participants With Modified Rankin Scale (0 - 1)
Description: Measures the degree of disability or dependence in the daily activities. Minimum score = 0 (best outcome - No symptoms); Maximum Score = 6 (worse outcome - dead)
Time Frame: 90 Days from Stroke Onset
Measure: Number; unit: percentage of participants
Arm/Group | Sham Transcranial Laser Therapy | Transcranial Laser Therapy
Number analyzed (Participants) | 7 | 5
percentage of participants | 42.9 | 40.0

ADVERSE EVENTS:
Arm/Group | Sham Transcranial Laser Therapy | Transcranial Laser Therapy
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/5
Other Adverse Events (participants affected / at risk) | 6/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Transcranial Laser Therapy (N=7) | Transcranial Laser Therapy (N=5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Clostridium colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Transcranial Laser Therapy (N=7) | Transcranial Laser Therapy (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Consitpation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1)
Ubiquinone decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrtion (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 2 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to device sponsor filing bankruptcy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No